CLINICAL TRIAL: NCT02605122
Title: A Phase 2/3, Randomized, Open-Label, Multi-center Study to Determine the Safety and Efficacy of Solithromycin in Adolescents and Children With Suspected or Confirmed Community-Acquired Bacterial Pneumonia
Brief Title: Safety and Efficacy of Solithromycin in Adolescents and Children With Community-Acquired Bacterial Pneumonia
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Development not proceeding
Sponsor: Melinta Therapeutics, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CE01-203
Record Dates: First submitted 2015-11-10; First posted 2015-11-16 (Estimated); Results first posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-11

CONDITIONS: Community-acquired Bacterial Pneumonia
Keywords: pneumonia; macrolide; pediatric
MeSH Terms: conditions — Pneumonia | interventions — solithromycin; Standard of Care; Ceftriaxone; Ampicillin; Amoxicillin; Amoxicillin-Potassium Clavulanate Combination; Azithromycin; Erythromycin; erythromycin lactobionate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A healthcare provider designated as a sub-investigator blinded to treatment allocation at the site documented clinical response at specified time points during the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Solithromycin (Experimental): Solithromycin will be administered orally, as capsules or as a suspension, or intravenously. Patients may receive intravenous therapy initially and switch to an oral formulation. Dosage is weight based and age based.
  Interventions: Drug: Solithromycin
- Standard of Care (Active Comparator): Comparators will be selected according to subject age and are consistent with current recommendations for treatment of CABP in children. These include intravenous ceftriaxone, ampicillin, and amoxicillin and oral amoxicillin and amoxicillin-clavulanic acid. Azithromycin or erythromycin may be added as well.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Solithromycin
  Other Names: CEM-101
  Arms: Solithromycin
Drug: Standard of Care — Age- and weight-based dosing as appropriate per sites standard of care.
  Other Names: ceftriaxone; ampicillin; amoxicillin; amoxicillin-clavulanic acid; Azithromycin; Erythromycin; Erythromycin lactobionate
  Arms: Standard of Care

SUMMARY:
This is a phase 2/3, randomized, open-label, active control, multi-center study to assess the safety and efficacy of solithromycin in children and adolescents with community-acquired bacterial pneumonia (CABP).

DETAILED DESCRIPTION:
Subjects who meet all inclusion/exclusion criteria and sign the informed consent/assent were enrolled. Subjects were randomized to receive solithromycin or a comparator antibiotic, administered IV and/or by mouth (PO) based on weight and age. Subjects were treated daily for 5 to 7 days with oral solithromycin and 5 to 7 days with IV or IV-to-oral solithromycin. Subjects were treated for 5 to 10 days with comparator antibiotics. Subjects received safety and efficacy assessments during and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* History of and/or documented fever (rectal, ear, or oral temperature ≥38°C or axillary temperature ≥37.5°C) or hypothermia (rectal, ear, or oral temperature <35°C or axillary temperature <34.5°C)
* Chest radiograph infiltrates consistent with bacterial pneumonia (or pneumonia caused by atypical bacterial agents); if a subject is outpatient and starting on oral therapy, a radiograph is not required.
* Presence of at least 2 of the following signs or symptoms:
* Cough
* Difficulty breathing
* Production of purulent sputum
* Chest pain
* Grunting
* Hypotension
* Tachycardia, defined as follows:

  2 months to <24 months: ≥160 beats/min 24 months to <10 years: ≥140 beats/min
  * 10 years: ≥100 beats/min
* Tachypnea, defined as follows:

  2 months to <12 months: ≥50 breaths/min 12 months to <5 years: ≥40 breaths/min
  * 5 years: ≥20 breaths/min
* Physical exam consistent with pulmonary consolidation
* Presence of at least 1 of the following:
* Leukocytosis (≥12,000 white blood cells [WBC]/mm3)
* Leukopenia (<5000 WBC/mm3)
* ≥10% immature neutrophils (bands) regardless of total peripheral WBC
* Elevated inflammatory markers (C-reactive protein or procalcitonin)
* Oxygen saturation <97% on room air
* Organism consistent with a typical respiratory pathogen identified

Exclusion Criteria:

* Ventilator-associated or hospital-acquired pneumonia
* >48 hours of systemic antibacterial therapy
* confirmed or suspected bacterial meningitis
* breast-feeding females
* positive pregnancy test

Ages: 2 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 97 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cohen-Wolkowiez, MD, PhD, Principal Investigator — Duke Clinical Research Institute
Locations (50):
- United States (21):
  - Little Rock, Arkansas
  - Los Angeles, California
  - Sacramento, California
  - San Diego, California
  - Washington D.C., District of Columbia
  - Tampa, Florida
  - Louisville, Kentucky
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - Durham, North Carolina
  - Greenville, North Carolina
  - Toledo, Ohio
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Memphis, Tennessee
  - Amarillo, Texas
  - Houston, Texas
  - Splendora, Texas
  - Charlottesville, Virginia
  - Richmond, Virginia
  - Roanoke, Virginia
- Bulgaria (5):
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Vratsa
- Hungary (12):
  - Budapest
  - Cegléd
  - Debrecen
  - Győr
  - Gyula
  - Mosdós
  - Nagykanizsa
  - Nyíregyháza
  - Szeged
  - Székesfehérvár
  - Törökbálint
  - Veszprém
- Philippines (7):
  - Caloocan
  - Cebu City
  - City of Muntinlupa
  - Davao City
  - Iloilo City
  - Manila
  - Quezon City
- Spain (4):
  - Esplugues de Llobregat, Barcelona
  - Donostia / San Sebastian, Guipuzcoa
  - Barcelona
  - Madrid
- London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects who met all inclusion/exclusion criteria and sign the informed consent/assent were enrolled. Subjects were randomized to receive solithromycin or a comparator antibiotic, administered IV and/or by mouth (PO) based on weight and age. Subjects received safety and efficacy assessments during and after treatment.
Groups:
- Solithromycin: Solithromycin was dosed for 5-7 days. Orally, as capsules or as a suspension, or intravenously. Subjects could receive intravenous therapy initially and switch to an oral formulation.
- Standard of Care: Comparators were dosed according to age and were consistent with current recommendations for treatment of CABP in children per site standard of care.
Period: Overall Study
Arm/Group | Solithromycin | Standard of Care
Started | 73 | 24
Received Study Drug | 70 | 24
Completed | 68 | 22
Not Completed | 5 | 2
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who receive at least one dose of study drug (solithromycin or active comparator) were included in the analysis population.
Groups:
- Solithromycin: Solithromycin was dosed for 5-7 days.
- Standard of Care: Comparators were does up to 10 days per site standard of care.
- Total: Total of all reporting groups
Arm/Group | Solithromycin | Standard of Care | Total
Number analyzed (Participants) | 70 | 24 | 94
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 70 | 24 | 94
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.48 (4.71) | 9.65 (4.95) | 9.57 (4.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 11 | 41
  Male | 40 | 13 | 53
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 65 | 21 | 86
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 4 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 2 | 13
  White | 47 | 16 | 63
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Hungary | 19 | 4 | 23
  United States | 18 | 9 | 27
  Philippines | 12 | 4 | 16
  Bulgaria | 21 | 6 | 27
  Spain | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overview of Adverse Events By Treatment Arm
Description: Summary of subjects experiencing Treatment Emergent Adverse Events (TEAE) through Day 16 visit and Treatment Emergent Serious Adverse Events (TESAE) through Day 28 visit (28 days +/- 4 days after randomization)
Time Frame: Up to 28 days post-treatment
Population: Treatment through Day 28 (28 days +/- 4days after randomization)
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care: Comparators were dosed up to 10 days per site standard of care.
Arm/Group | Solithromycin | Standard of Care
Number analyzed (Participants) | 70 | 24
Participants
  TEAE | 24 | 7
  TESAE | 1 | 1
Statistical Analysis 1: Comparison: Solithromycin vs Standard of Care; Test type: Other; Clopper-Pearson — No p-value was performed. Study prematurely discontinued. Clopper-Pearson analysis was used to determine confidence intervals; Proportion experiencing TEAE or TESAE = 34.3, 95% CI 2-sided [23 to 47]

2. Secondary Outcome: Summary of Early Clinical Response
Description: Early clinical response (ECR) was defined using the latest efficacy evaluation from Day 2 (if subject discharged prior to Day 2), Day3, or Day 4, and was defined as improvement in at least 1 presenting sign/symptom of CABP with no deterioration in any signs/symptoms of CABP and no requirement for an additional antibiotic.
Time Frame: During Treatment Days 3 to 4
Population: Not all subjects had the Early Clinical Improvement assessment performed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Solithromycin | Standard of Care
Number analyzed (Participants) | 51 | 15
percentage of participants | 66.7 [52 to 79] | 46.7 [21 to 73]
Statistical Analysis 1: Comparison: Solithromycin vs Standard of Care; Test type: Other; Clopper-Pearson — [p-value comment as in outcome 1, analysis 1]; Achievement of ECR = 62.1, 95% CI 2-sided [49 to 74]

3. Secondary Outcome: Summary of Clinical Improvement
Description: Clinical improvement was assessed using the latest efficacy evaluation conducted on last day of treatment (+48 hours), and was defined identically to the early clinical response.
Time Frame: Last day of Treatment (+48 hours)
Population: Not all subjects had the Clinical Improvement assessment performed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Solithromycin | Standard of Care
Number analyzed (Participants) | 62 | 21
percentage of participants | 64.5 [51 to 76] | 81 [58 to 95]
Statistical Analysis 1: Comparison: Solithromycin vs Standard of Care; Test type: Other; Clopper-Pearson — [p-value comment as in outcome 1, analysis 1]; Achievement of Clinical Improvement = 68.7, 95% CI 2-sided [58 to 78]

4. Secondary Outcome: Summary of Clinical Cure
Description: Clinical cure was assessed using the latest efficacy evaluation conducted on Day 16 (+/- 4 days) post-randomization, and was defined as resolution of all presenting signs/symptoms of CABP (excluding cough), no development of new signs/symptoms of CABP, and no requirement for an additional antibiotic.
Time Frame: Short-term follow-up at 16 days (+/- 4 days)
Population: Not all subjects had the Clinical cure assessment performed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Solithromycin | Standard of Care
Number analyzed (Participants) | 60 | 19
percentage of participants | 60.0 [47 to 72] | 68.4 [43 to 87]
Statistical Analysis 1: Comparison: Solithromycin vs Standard of Care; Test type: Other; Clopper-Pearson — No p-value was performed. Study prematurely discontinued. Clopper-Pearson was used to determine confidence intervals; Achievement of Clinical Cure = 62, 95% CI 2-sided [50 to 73]

ADVERSE EVENTS:
Time Frame: Up to 32 days
Groups:
- Standard of Care: Comparators were dosed up to 10 days per sites standard of care.
Arm/Group | Solithromycin | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/70 | 1/24
Other Adverse Events (participants affected / at risk) | 24/70 | 7/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solithromycin (N=70) | Standard of Care (N=24)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Viral (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Solithromycin (N=70) | Standard of Care (N=24)
Phlebitis (Vascular disorders) | 5 (5) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 3 (3) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 0 (0)
Oxygen Saturation Decreased (Investigations) | 1 (1) | 0 (0)
Transaminases Increased (Investigations) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Infusion Site Pain (General disorders) | 6 (6) | 0 (0)
Infusion Site Pruritus (General disorders) | 1 (1) | 0 (0)
Infusion Site Urticaria (General disorders) | 1 (1) | 0 (0)
Injection Site Reaction (General disorders) | 1 (1) | 0 (0)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (4)
Abdominal Discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Infectious Pleural Effusion (Infections and infestations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was discontinued early due to a company business decision. Study discontinuation was not related to safety or tolerability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study Site will not submit its results for independent publication until after a coordinated, multicenter Study publication has been submitted or one (1) year after the conclusion of the Study, whichever occurs first. Study Site and/or Investigator shall submit any proposed publication or presentation resulting from Study Site's performance of the Protocol to the Prime Recipient for review and comment at least forty-five (45) days prior to the date of submission.

DOCUMENTS (2):
  • Study Protocol (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT02605122/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/22/NCT02605122/SAP_001.pdf